CLINICAL TRIAL: NCT00451425
Title: Weight Gain During Pregnancy - a Randomized Controlled Trial of Intervention to Prevent Excessive Gestational Weight Gain.
Acronym: VIGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Modrahalsovard Orebro lan, Orebro lans landsting
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 2007/031
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Weight Gain
Keywords: pregnancy; weight gain; obesity; macrosomia
MeSH Terms: conditions — Weight Gain; Obesity | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- control (No Intervention): standard maternity care
  Interventions: Behavioral: motivational intervention in pregnancy

INTERVENTIONS:
Behavioral: motivational intervention in pregnancy — Motivational program including individualized counseling on diet and physical activity

SUMMARY:
Excessive weight gain during pregnancy is associated with complications during delivery primarily due to macrosomia (large babies) but also with high levels of weight retention post pregnancy and thereby increased risk of future weight related health problems. The primary aim of this study is to evaluate the efficacy of an intervention consisting of; recurrent Motivational Interviewing (MI), prescription of physical activity and extended information on recommended weight gain during pregnancy in regards to preventing excessive gestational weight gain.

ELIGIBILITY:
Inclusion Criteria:

* >18 years,
* Adequate language skills (swedish),
* BMI>19.9,
* Pregnancy estimated <16 weeks (LMP),
* Planned for basic pregnancy surveillance (healthy mother).

Exclusion Criteria:

* History of eating disorder,
* History of having a growth restricted child.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The number of women with a weight gain during pregnancy within IOM´s recommendation is compared between study groups. | 9 months

SECONDARY OUTCOMES:
Weight retention(kg) up until one year after delivery is compared between study groups. | one year after delivery
Number of fetal and maternal complications in pregnancy is compared between study groups | 9 months
Number of fetal and maternal complications during delivery is compared between study groups | during delivery
Child birth weight and weight development of the child up to one year of age is compared between study groups. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Nilsson, MD. MD, Study Chair — Region Örebro County
Locations (1):
- Modrahalsovarden Orebro lan, Örebro, Sweden

REFERENCES:
- [Derived] Ronnberg AK, Ostlund I, Fadl H, Gottvall T, Nilsson K. Intervention during pregnancy to reduce excessive gestational weight gain-a randomised controlled trial. BJOG. 2015 Mar;122(4):537-44. doi: 10.1111/1471-0528.13131. Epub 2014 Nov 4. PMID 25367823